CLINICAL TRIAL: NCT03509259
Title: Discovering Risk Factors for Cardiovascular Diseases in Elderly Asthma
Brief Title: Cardiovascular Diseases in Elderly Asthma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: L-2017-313
Record Dates: First submitted 2018-03-29; First posted 2018-04-26 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma: If the doctor has been diagnosed with asthma and one or more of the following criteria is met;
  1. FEV1 (Forced expiratory volume in 1 second) increased more than 12% & 200 mL after 10-20 minutes of inhalation of short-acting bronchodilator (200-400 mg salbutamol)
  2. Positive bronchial provocation tests (methacholine, mannitol, exercise, aspirin, etc.)
  3. FEV1 Increased more than 12% & 200 mL from baseline FEV1 after anti-inflammatory treatment for 4 weeks or longer.
  They can have concomittent COPD or not
- Healthy control: Subjects who performed coronary artery calcium scoring CT for health checkup purpose.(retrospective group = historical control group)

SUMMARY:
This study is a cross-sectional study to evaluate the relationship between coronary calcium score and clinical parameters of asthma such as onset of disease, lung function parameter and airway inflammation parameter (sputum eosinophil or FeNO) in Korean elderly asthma (regardless of whether they have concomittent COPD or not) patients

DETAILED DESCRIPTION:
Subjects who visited Allergy Clinic in SMG-SNU Boramae Medical Center for asthma or ACO will be recruited consecutively. Subjects who meets the inclusion criteria and agree to participate in the study will take coronary artery calcium scoring CT and asthma CT (inspiration and expiration images). The correlation between the degree of coronary calcification and airway diameter, airway wall thickness, air-trapping and emphysema will be evaluated as well as clinical parameters of asthma. We will also compare those correlations from the images of healthy control subjects who performed the coronary calcium scoring CT for health checkup purpose.

ELIGIBILITY:
Inclusion Criteria:

* If the doctor has been diagnosed with asthma and one or more of the following criteria is met;

  1. FEV1 increased more than 12% & 200 mL after 10-20 minutes of inhalation of short-acting bronchodilator (200-400 mg salbutamol)
  2. Positive bronchial provocation tests (methacholine, mannitol, exercise, aspirin, etc.)
  3. FEV1 Increased more than 12% & 200 mL from baseline FEV1 after anti-inflammatory treatment for 4 weeks or longer.

Exclusion Criteria:

* Those who were already diagnosed and treated for coronary artery diseases.
* Those with other structural lung diseases such as Tuberculosis destroyed lung and interstitial lung diseases
* Those who are unable to conduct a test or questionnaire due to severe systemic illness, or cognitive dysfunction.
* Those who are participating in other clinical trial using IND(investigational new drug) or finished other clinical trial within 30 days.
* Those who refuse to participate in the study or withdraw the consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who visited Allergy Clinic in SMG-SNU Boramae Medical Center for asthma or ACO
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
coronary calcium score | through study completion, an average of 1 month
  coronary calcium score from coronary calcium scoring CT which, we assumed to be a surrogate marker for cardiovascular risk.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Suk Yang, MD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided